CLINICAL TRIAL: NCT04531007
Title: Validation of Intravascular Imaging and Physiology for Intermediate Left Main Stem Stenosis With Downstream Coronary Lesions
Brief Title: Imaging and Physiology for Intermediate Left Main Stem Stenosis
Acronym: VIP-LMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Daniel Chamié, Principal Investigator, Instituto Dante Pazzanese de Cardiologia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4978/2019
Record Dates: First submitted 2020-06-26; First posted 2020-08-28 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Disease Left Main
Keywords: Left Main Coronary Artery (LMCA); FFR; iFR; OCT; IVUS; intracoronary imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermediate LMS stenosis (Experimental): Patients with intermediate left main stem stenosis with additional severe downstream lesion will be subject to physiology (FFR and iFR) at multiple sites along the target vessels before and after PCI of the severe lesion located in the downstream vessel. Intravascular imaging (IVUS and OCT) will be performed for additional evaluation of the left main stem stenosis.
  Interventions: Diagnostic Test: iFR/ FFR/ IVUS/ OCT

INTERVENTIONS:
Diagnostic Test: iFR/ FFR/ IVUS/ OCT — intermediate lesion evaluation with intracoronary physiology and imaging

SUMMARY:
The present research aims to determine the impact of stenoses in downstream vessels on the FFR and iFR measurements of left main coronary artery (LMCA) stenoses of intermediate severity as determined by coronary angiography. Anatomic metrics derived from intravascular imaging modalities of IVUS and optical coherence tomography (OCT) will also be validated using as the comparator the FFRtrue and iFRtrue measurements pf LMCA lesions.

DETAILED DESCRIPTION:
Accurate characterization of the functional significance of intermediate stenoses located in the left main coronary artery (LMCA) is of central relevance for decisions about the need of myocardial revascularization. However, the physiological assessment of such lesions by means of fractional flow reserve (FFR) measurements are affected by stenoses in the downstream vessels (left anterior descending artery and/or left circumflex artery), which frequently coexist in series with LMCA lesions. More recently introduced, the instantaneous wave-free ratio (iFR) is a resting index that is less influenced by crosstalk between serial lesions and, in theory, could be more accurate for assessment of LMCA stenoses in the presence of downstream disease. Nonetheless, iFR has not been validated for assessment of LMCA lesions. Due to the difficulty in interpreting FFR results, the possibility of characterizing the atheroma type, precisely estimate lesion severity and disease extension and distribution, intravascular imaging [especially intravascular ultrasound (IVUS)] became an attractive alternative to assess LMCA lesions and guide the percutaneous treatment, whenever this strategy is selected. However, most IVUS validations for LMCA stenosis assessment used FFR as the standard comparator, which by itself has limited diagnostic ability in this anatomic scenario.

Thus, the main objective of the current research project is to determine the impact of stenoses in downstream vessels on FFR and iFR measurements of LMCA stenoses of intermediate severity as determined by coronary angiography. The primary endpoint is the change (delta) in FFR and iFR values prior and after percutaneous treatment of downstream stenoses. Assuming a change of 0.04 mmHg between the FFRpredicted and FFRtrue with a standard deviation of 0.04 mmHg, and a change of 0.01 mmHg between iFRpredicted and iFRtrue with a standard deviation of 0.03 mmHg, a total of 53 patients are needed to confirm the mean difference of 0.03 mmHg between iFR and FFR changes before and after treatment of downstream stenoses. Anatomic metrics derived from intravascular imaging modalities of IVUS and optical coherence tomography (OCT) will also be validated using as the comparator the FFRtrue and iFRtrue measurements.

ELIGIBILITY:
Inclusion Criteria:

- age >/= 18 years;

* patients who have an intermediate (40-70% diameter stenosis) lesion located in the LMS and a concomitant significant (>/=70% diameter stenosis) in one of the two major downstream vessels (the LAD or the LCx). The severity of LMS and downstream lesions will be assessed by visual estimation of the coronary angiography;
* need of complementary diagnostic work up to ascertain the functional/physiological significance of the LMS lesion, that is not possible from the analysis of angiographic images only:

  * Intermediate severity of LMS lesion, or angiographic ambiguity;
  * Impossibility to conclusively associate the LMS lesion with the patient's symptoms/clinical presentation due to confounders introduced by the significant downstream lesion;
  * Impossibility to conclusively determine the severity and functional/physiological significance of the LMS lesion solely by the visual analysis of the coronary angiography;
  * Impossibility to conclusively determine the relative contribution of the LMS lesion to the ischemic burden determined by non-invasive functional tests due to the presence of a significant downstream lesion;
* Clinical indication for PCI of the downstream lesion located in the LAD or LCx:

  * stable angina unresponsive to optimized medical treatment;
  * important ischemic burden (> 10% of myocardial mass in territories supplied by the diseased vessels);
  * Reduced FFR/iFR values indicative of myocardial ischemia with significant pressure gradient across the downstream lesion;
  * Acute coronary syndrome without ST elevation or stabilized (>7 days) acute myocardial infarction;
* Downstream lesion anatomically suited for PCI;
* LMS anatomy suited for PCI, with a low or intermediate SYNTAX score (< 32);
* Lack of contra-indications for second-generation drug-eluting stents and/or use of dual antiplatelet therapy for at least 6 months.

Exclusion Criteria:

Left ventricular ejection fraction £ 40%;

* Renal dysfunction with a glomerular filtration rate £ 45 mL/min;
* Concomitance of right coronary artery occlusion supplied by collateral circulation from the left coronary;
* Prior coronary artery bypass graft with at least on patent graft to any vessel of the left coronary;
* Concomitant significant valvular heart disease;
* The first 7 days of an acute myocardial infarction;
* Downstream lesion located only in branches from the major downstream vessels (e.g. diagonal branches of LAD or obtuse marginal branches of the LCx);
* Downstream lesions located in the distal segments of LAD or LCx;
* Significant tortuosity of the downstream vessels in which difficulty to navigate with the physiology wire and/or intravascular imaging catheter is anticipated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of iFR and FFR values of the LMS stenosis before and after PCI of the significant downstream stenosis | diagnostic procedure
  determine the change of iFR and FFR values of the LMS stenosis before and after PCI of the significant downstream stenosis (iFRtrue - iFRpred and FFRtrue - FFRpred)
Accuracy of intravascular imaging in predicting functionally signifcant LMS stenosis | diagnostic procedure
  establish the diagnostic accuracy of the minimum lumen areas determined by IVUS and OCT in the LMS in comparison with the iFRtrue and FFRtrue)

SECONDARY OUTCOMES:
Accuracy of pressure changes in the iFR and FFR pullback curves before PCI of the downstream lesion in predicting the functional significance of LMS stenosis | diagnostic procedure
  Establish the accuracy of pressure changes in the iFR and FFR pullback curves before PCI of the downstream lesion to predict the iFRtue and FFRtrue observed after PCI of the downstream lesion;
Accuracy of iFRpred-contra and FFRpred-contra before PCI of the downstream lesion in predicting the functional significance of LMS stenosis | diagnostic procedure
  Establish the ability of iFRpred-contra and FFRpred-contra before PCI of the downstream lesion in predict the iFRtrue and FFRtrue of the LMS stenosis;
Agreement of the iFRcontra and FFRcontra after PCI of the downstream stenosis with the iFRtrue and FFRtrue. | diagnostic procedure
  Verify the agreement of the iFRcontra and FFRcontra after PCI of the downstream stenosis with the iFRtrue and FFRtrue.
Accuracy of minimum lumen area determined by IVUS and OCT in the LMS to predict the functional significance of LMS stenosis | diagnostic procedure
  Diagnostic accuracy of the minimum lumen area in the LMS by IVUS and OCT to predict iFRtrue and FFRtrue of the LMS stenosis
Accuracy of minimum lumen diameter determined by IVUS and OCT in the LMS to predict the functional significance of LMS stenosis | diagnostic procedure
  Diagnostic accuracy of the minimum lumen diameter in the LMS by IVUS and OCT to predict iFRtrue and FFRtrue of the LMS stenosis
Accuracy of percent diameter stenosis determined by IVUS and OCT in the LMS to predict the functional significance of LMS stenosis | diagnostic procedure
  Diagnostic accuracy of the percent diameter stenosis in the LMS by IVUS and OCT to predict iFRtrue and FFRtrue of the LMS stenosis
Accuracy of percent area stenosis determined by IVUS and OCT in the LMS to predict the functional significance of LMS stenosis | diagnostic procedure
  Diagnostic accuracy of the percent area stenosis in the LMS by IVUS and OCT to predict iFRtrue and FFRtrue of the LMS stenosis
Accuracy of lesion length determined by IVUS and OCT in the LMS to predict the functional significance of LMS stenosis | diagnostic procedure
  Diagnostic accuracy of lesion length in the LMS by IVUS and OCT to predict iFRtrue and FFRtrue of the LMS stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chamie, MD, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Fausto Feres, MD, PhD, Study Chair — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No